CLINICAL TRIAL: NCT04343963
Title: Pyridostigmine in Patients With Severe Acute Respiratory Syndrome Secondary to SARS-CoV-2 Infection
Brief Title: Pyridostigmine in Severe SARS-CoV-2 Infection
Acronym: PISCO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inf-3323
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Pyridostigmine Bromide; Starch

STUDY DESIGN:
Intervention Model Description: Participants will receive pyridostigmine at a dose of 60 mg / day (or matching placebo), P.O. during a period of up to 14 days, until hospital discharge, death, mechanical ventilation, or increase in the SOFA scale ≥2 points.
  The proposed dose is a safe dose according to the experience in myasthenia gravis and healthy people, as well as in at least three clinical studies in people living with HIV.
  Participants will be double-blind 1: 1 randomized to receive pyridostigmine or placebo for up to 14 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyridostigmine (Active Comparator): Pyridostigmine bromide tablet (60mg P.O. once per day for 14 days)
  Interventions: Drug: Pyridostigmine Bromide
- Placebo (Placebo Comparator): Placebo tablet (60mg P.O. once per day for 14 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine Bromide — One 60mg tablet P.O. once per day for 14 days
  Other Names: Mestinon; Pyridostigmine
  Arms: Pyridostigmine
Drug: Placebo — One tablet P.O. once per day for 14 days
  Other Names: Starch (pharmaceutical grade)
  Arms: Placebo

SUMMARY:
We will evaluate low-dose pyridostigmine as add-on therapy to best medical care in patients with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection and its related Coronavirus Disease 2019 (COVID-19) who require hospitalization. Our hypothesis is that, in comparison to the placebo, pyridostigmine will reduce in at least 10% a composite outcome [death; mechanical ventilation; >2 point-increase in the SOFA score) by day 28. We will also evaluate interleukin (IL)-6 kinetics during the first 14 days of in-hospital stay.

It is estimated that 25-33% of patients hospitalized for COVID-19 are admitted to intensive care units (ICU) for severe hypoxemia. The reported mortality in those with severe disease ranges between 38% and 49%. So far, there is no pharmacological therapeutic (or else) strategy known to reduce morbidity and mortality in these patients. Mortality in COVID-19 appears to be mediated not necessarily by the direct effect of the infection, but by the disproportionate inflammatory response of the host.

Pyridostigmine is an old drug that, by inhibiting acetylcholine-esterase, the enzymatic machinery that degrades acetylcholine (ACh), results in increased ACh bioavailability. ACh, in turn, ligates to nicotinic-alpha7 receptors in macrophages and T cells, resulting in reduced overactivation of these immune cells. In experimental murine sepsis, this family of drugs has resulted in reduced inflammation and mortality. Human evidence is scarce for severe inflammatory conditions. However, recent evidence from our group and others indicates that pyridostigmine has an immunomodulatory effect in people living with HIV, resulting in elevation of CD4+ T cell counts, decreased immune activation, and reduction in inflammatory mediators. Altogether, this suggests that ACh-esterase inhibitors may act as immunomodulators during viral infections, potentially reducing the inflammatory cascade (the so-called "cytokine storm") observed in critically ill COVID-19 patients.

At the proposed dose (60mg/d), the rate of minor adverse events is less than 5% with no reported serious adverse effects. From that perspective, we consider that pyridostigmine can function as an immuno-modulator and reduce morbidity and mortality in COVID-19-stricken patients, with the added value of a safe pharmacological profile. Moreover, as an old drug, re-purposing it for a novel indication may be a simpler, more efficient approach than developing a novel one from the ground up.

DETAILED DESCRIPTION:
The study will be divided into two phases, each with different variables to evaluate, as described below:

The primary objective of the first phase (proof-of-concept) will be to evaluate the effect of pyridostigmine on the serum level of interleukin (IL)-6 as an indicator of severe inflammation, as well as its kinetics throughout the days that the patient is hospitalized.

In the first phase, we will evaluate the safety and feasibility of the study in a representative sample and we will explore in a preliminary way the magnitude of the effect of the intervention. Safety will be evaluated according to the adverse effects reported in patients with acute intoxication (accidental or in suicide attempt) with pyridostigmine:

1. Abdominal pain/cramps
2. Diarrhea
3. Vomiting, nausea, or both
4. Hypersalivation
5. Urinary incontinence
6. Fasciculations or muscle weakness
7. Blurred vision

In the second phase (to be carried out only if the results of the first phase justify it), the primary outcome to be evaluated is mortality, the requirement of invasive or non-invasive mechanical ventilation, or an increase in the SOFA scale ≥2 points.

The following secondary outcomes were evaluated: changes in the total SOFA score between study entry and evaluation at 3, 7, and 14 days; the number of days of hospital stay, days of hospitalization in the intensive care unit, and the need (and if applicable, the number of days required) for invasive or non-invasive mechanical ventilation.

The variables to measure are sex, age at hospitalization, date of COVID-19 diagnosis, date and SOFA scale measurement, date of hospitalization, date of transfer to the intensive care unit, date of initiation of mechanical ventilation. , date and reason for leaving the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old)
2. Signed informed consent by the patient or designated legal representative
3. Confirmatory laboratory test for SARS-CoV-2 / COVID-19 infection
4. Pneumonia confirmed by imaging studies
5. Agree to venous blood collection according to the protocol
6. Need for hospitalization with increased mortality criteria according to published observations, including one or more of the following severity criteria according to the treating medical team:

   * a. Dyspnoea
   * b. Lung infiltrates> 50% of lung fields by CT
   * c. A ratio of partial pressure arterial oxygen (PaO2) to the fraction of inspired oxygen (FiO2) <300 mmHg
   * d. Pulse oximetry <90% to ambient air, or a 3% drop in baseline oximetry, or need to increase supplemental oxygen due to chronic hypoxia, as well as the need for supplemental oxygen according to medical judgment

And, alteration of one or more of the following laboratory studies at the time of hospital admission:

* i. D-dimer >1 ug/mL
* ii. Ferritin level >300 ng/mL
* iii. C-reactive protein (CRP) >3mg/L
* iv. Lactate dehydrogenase (LDH) >245 U/L
* v. Lymphopenia <800 cells/uL
* vi. Creatine kinase (CK) level >800 IU/L

Exclusion Criteria:

1. Pyridostigmine allergy
2. If female, pregnancy or breastfeeding
3. Meet the following critical illness criteria before signing informed consent and taking the first dose of study medication:

   1. . Need for mechanical ventilation
   2. . Admission to the ICU for any reason
   3. . Meet criteria for sepsis or septic shock
4. Concomitant autoimmune diseases
5. Known immunodeficiency (including HIV infection)
6. Need for mechanical ventilation before signing informed consent and taking the first dose of study medication
7. Inability to administer orally / enterally
8. Use of immunosuppressants or immuno-modulators in the preceding 28 days, including chemotherapeutics and steroids, unless recommended by the treatment medical team as part of the therapeutic approach for SARS-CoV-2 infection
9. Participation in interventional clinical trials in the preceding 28 days (however, participation in observational trials or those with no therapeutic intervention, is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Critical condition or death | 28 days
  Composite of death, Need for mechanical ventilation, or an increase of 2 or more points in the SOFA score
IL-6 | 14 days in-hospital, hospital discharge, or death
  Kinetics of circulating IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Sergio I Valdés-Ferrer, MD, PhD, Study Chair — Instituto Nacional De Ciencias Médicas y Nutrición
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Chavan SS, Tracey KJ. Essential Neuroscience in Immunology. J Immunol. 2017 May 1;198(9):3389-3397. doi: 10.4049/jimmunol.1601613. PMID 28416717
- [Background] Koopman FA, Chavan SS, Miljko S, Grazio S, Sokolovic S, Schuurman PR, Mehta AD, Levine YA, Faltys M, Zitnik R, Tracey KJ, Tak PP. Vagus nerve stimulation inhibits cytokine production and attenuates disease severity in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2016 Jul 19;113(29):8284-9. doi: 10.1073/pnas.1605635113. Epub 2016 Jul 5. PMID 27382171
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Rosas-Ballina M, Valdes-Ferrer SI, Dancho ME, Ochani M, Katz D, Cheng KF, Olofsson PS, Chavan SS, Al-Abed Y, Tracey KJ, Pavlov VA. Xanomeline suppresses excessive pro-inflammatory cytokine responses through neural signal-mediated pathways and improves survival in lethal inflammation. Brain Behav Immun. 2015 Feb;44:19-27. doi: 10.1016/j.bbi.2014.07.010. Epub 2014 Jul 23. PMID 25063706
- [Background] Valdes-Ferrer SI, Crispin JC, Belaunzaran PF, Cantu-Brito CG, Sierra-Madero J, Alcocer-Varela J. Acetylcholine-esterase inhibitor pyridostigmine decreases T cell overactivation in patients infected by HIV. AIDS Res Hum Retroviruses. 2009 Aug;25(8):749-55. doi: 10.1089/aid.2008.0257. PMID 19645607
- [Background] Robinson-Papp J, Nmashie A, Pedowitz E, George MC, Sharma S, Murray J, Benn EKT, Lawrence SA, Machac J, Heiba S, Kim-Schulze S, Navis A, Roland BC, Morgello S. The effect of pyridostigmine on small intestinal bacterial overgrowth (SIBO) and plasma inflammatory biomarkers in HIV-associated autonomic neuropathies. J Neurovirol. 2019 Aug;25(4):551-559. doi: 10.1007/s13365-019-00756-9. Epub 2019 May 16. PMID 31098925
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Derived] Fragoso-Saavedra S, Nunez I, Audelo-Cruz BM, Arias-Martinez S, Manzur-Sandoval D, Quintero-Villegas A, Benjamin Garcia-Gonzalez H, Carbajal-Morelos SL, PoncedeLeon-Rosales S, Gotes-Palazuelos J, Maza-Larrea JA, Rosales-de la Rosa JJ, Diaz-Rivera D, Luna-Garcia E, Piten-Isidro E, Del Rio-Estrada PM, Fragoso-Saavedra M, Caro-Vega Y, Batina I, Islas-Weinstein L, Iruegas-Nunez DA, Calva JJ, Belaunzaran-Zamudio PF, Sierra-Madero J, Crispin JC, Valdes-Ferrer SI. Pyridostigmine reduces mortality of patients with severe SARS-CoV-2 infection: A phase 2/3 randomized controlled trial. Mol Med. 2022 Nov 8;28(1):131. doi: 10.1186/s10020-022-00553-x. PMID 36348276
- [Derived] Fragoso-Saavedra S, Iruegas-Nunez DA, Quintero-Villegas A, Garcia-Gonzalez HB, Nunez I, Carbajal-Morelos SL, Audelo-Cruz BM, Arias-Martinez S, Caro-Vega Y, Calva JJ, Luqueno-Martinez V, Gonzalez-Duarte A, Crabtree-Ramirez B, Crispin JC, Sierra-Madero J, Belaunzaran-Zamudio PF, Valdes-Ferrer SI. A parallel-group, multicenter randomized, double-blinded, placebo-controlled, phase 2/3, clinical trial to test the efficacy of pyridostigmine bromide at low doses to reduce mortality or invasive mechanical ventilation in adults with severe SARS-CoV-2 infection: the Pyridostigmine In Severe COvid-19 (PISCO) trial protocol. BMC Infect Dis. 2020 Oct 16;20(1):765. doi: 10.1186/s12879-020-05485-7. PMID 33066761